CLINICAL TRIAL: NCT02030405
Title: A Phase 2 Study of Single-Agent MLN9708 for the Treatment of Relapsed or Refractory Acute Myeloid Leukemia With Mutated Nucleophosmin-1
Brief Title: Ixazomib (MLN9708) in Treating Patients With Relapsed or Refractory Acute Myeloid Leukemia
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Regulatory
Sponsor: Steven E. Coutre (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor-Investigator, Steven E. Coutre, Assistant Professor of Medicine, Stanford University
Organization: Stanford University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-28771; NCI-2013-02231 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); P30CA124435 (NIH); HEMAML0028 (Other: OnCore Number)
Record Dates: First submitted 2013-11-25; First posted 2014-01-08 (Estimated); Results first posted 2017-03-10 (Actual); Last update posted 2019-04-05 (Actual); Status verified 2019-04

CONDITIONS: Adult Acute Megakaryoblastic Leukemia (M7); Adult Acute Minimally Differentiated Myeloid Leukemia (M0); Adult Acute Monoblastic Leukemia (M5a); Adult Acute Monocytic Leukemia (M5b); Adult Acute Myeloblastic Leukemia With Maturation (M2); Adult Acute Myeloblastic Leukemia Without Maturation (M1); Adult Acute Myeloid Leukemia With 11q23 (MLL) Abnormalities; Adult Acute Myeloid Leukemia With Del(5q); Adult Acute Myeloid Leukemia With Inv(16)(p13;q22); Adult Acute Myeloid Leukemia With t(16;16)(p13;q22); Adult Acute Myeloid Leukemia With t(8;21)(q22;q22); Adult Acute Myelomonocytic Leukemia (M4); Adult Erythroleukemia (M6a); Adult Pure Erythroid Leukemia (M6b); Recurrent Adult Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Megakaryoblastic, Acute; Leukemia, Monocytic, Acute; Leukemia, Myeloid, Acute; Congenital Abnormalities; Leukemia, Myelomonocytic, Acute; Leukemia, Erythroblastic, Acute | interventions — ixazomib; Proteasome Inhibitors

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Ixazomib (MLN9708) (Experimental): Participants receive ixazomib PO (orally) on days 1, 4, 8, and 11. Treatment repeats every 21 days for up to 12 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Ixazomib

INTERVENTIONS:
Drug: Ixazomib — Given orally (PO)
  Other Names: Ninlaro; MLN9708; proteasome inhibitor

SUMMARY:
This phase 2 trial studies how well ixazomib(MLN9708) works in treating study participants with relapsed or refractory acute myeloid leukemia. Ixazomib may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

Determine the best response including complete remission (CR), CR with incomplete recovery (CRi), and partial remission (PR) after 3 cycles of treatment with MLN9708 (ixazomib) in participants with nucleophosmin (NPM)1-mutated acute myeloid leukemia (AML) (following the LeukemiaNet1 guidelines for response criteria).

SECONDARY OBJECTIVES:

* Determine the duration of remission in all responders after treatment with MLN9708 defined as the time of documented remission until relapse.
* Determine the 1 year overall survival, which will be measured from time of study entry to the earlier of death from any cause or end of follow up at 1 year.
* Establish toxicity and tolerability of MLN9708 treatment in AML, including non-hematologic toxicities grade 3 or above as specified by Common Terminology Criteria for Adverse Events (CTCAE) version 4.0.

OUTLINE:

Participants receive ixazomib orally (PO) on days 1, 4, 8, and 11. Treatment repeats every 21 days for up to 12 courses in the absence of disease progression or unacceptable toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of relapsed or refractory AML of any French American British (FAB) subtype except M3 and NPM1 genetic mutation detected by molecular assay; AML patients treated at Stanford have NPM1 molecular mutation status checked routinely at time of diagnosis in a Clinical Laboratory Improvement Amendment (CLIA)-certified laboratory
* Male or female patients and no race-ethnic restrictions
* Patients are unwilling, or who are determined to be medically unfit for or resistant to standard intensive induction chemotherapy; patients who are medically unfit will be determined by the treating primary hematologist and the principal investigator (including but not limited to evaluation of co-morbidities, and response and complications to previous AML treatment strategy)
* Eastern Cooperative Oncology Group (ECOG) 0 to 2
* Ability to understand and the willingness to sign a written informed consent document
* Female patients who:

  * Are postmenopausal for at least 1 year before the screening visit, OR
  * Are surgically sterile, OR
  * If they are of childbearing potential, agree to practice 2 effective methods of contraception, at the same time, from the time of signing the informed consent form through 90 days after the last dose of study drug, AND
  * Must also adhere to the guidelines of any treatment-specific pregnancy prevention program, if applicable, OR
  * Agree to practice true abstinence when this is in line with the preferred and usual lifestyle of the subject; (periodic abstinence [eg, calendar, ovulation, symptothermal, post-ovulation methods] and withdrawal are not acceptable methods of contraception)
* Male patients, even if surgically sterilized (ie, status post-vasectomy), must agree to one of the following:

  * Agree to practice effective barrier contraception during the entire study treatment period and through 90 days after the last dose of study drug, OR
  * Must also adhere to the guidelines of any treatment-specific pregnancy prevention program, if applicable, OR
  * Agree to practice true abstinence when this is in line with the preferred and usual lifestyle of the subject; (periodic abstinence (eg, calendar, ovulation, symptothermal, post-ovulation methods] and withdrawal are not acceptable methods of contraception)
* Total bilirubin ≤ 1.5 x the upper limit of the normal range (ULN)
* Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 3 x ULN
* Calculated creatinine clearance ≥ 30 mL/min

Exclusion Criteria:

* Female patient who are lactating or have a positive serum pregnancy test during the screening period
* Major surgery within 14 days before enrollment
* Radiotherapy within 14 days before enrollment; if the involved field is small, 7 days will be considered a sufficient interval between treatment and administration of MLN9708
* Known active and uncontrolled central nervous system (CNS) involvement of leukemia (a lumbar puncture does not need to be performed as a part of screening)
* Have a significant uncontrolled infection active infection
* Have other severe concurrent disease or serious organ dysfunction involving the heart, kidney, liver or other organ system that may place the patient at undue risk to undergo treatment including uncontrolled hypertension, uncontrolled cardiac arrhythmias, symptomatic congestive heart failure, unstable angina, or myocardial infarction within the past 6 months
* Systemic treatment, within 14 days before the first dose of MLN9708, with strong inhibitors of cytochrome P450, family 1, subfamily A, polypeptide 2 (CYP1A2) (fluvoxamine, enoxacin, ciprofloxacin), strong inhibitors of cytochrome P450, family 3, subfamily A (CYP3A) (clarithromycin, telithromycin, itraconazole, voriconazole, ketoconazole, nefazodone, posaconazole) or strong CYP3A inducers (rifampin, rifapentine, rifabutin, carbamazepine, phenytoin, phenobarbital), or use of Ginkgo biloba or St. John's wort
* Known ongoing or active systemic infection, active hepatitis B or C virus infection, or known human immunodeficiency virus (HIV) positive
* Known gastrointestinal (GI) disease or GI procedure that could interfere with the oral absorption or tolerance of MLN9708 including difficulty
* Diagnosed or treated for another malignancy within 2 years before study enrollment or previously diagnosed with another malignancy and have any evidence of residual disease; patients with nonmelanoma skin cancer or carcinoma in situ of any type are not excluded if they have undergone complete resection; this does not preclude previous diagnosis of acute myeloid leukemia or myelodysplastic syndrome
* Patient has ≥ grade 3 peripheral neuropathy, or grade 2 with pain on clinical examination during the screening
* Participation in other clinical trials, including those with other investigational agents not included in this trial, within 21 days of the start of this trial and throughout the duration of this trial
* Known allergy to any of the study medications, their analogues, or excipients in the various formulations of any agent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2014-03; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bruno de Medeiros, Principal Investigator — Stanford University Hospitals and Clinics
Locations (1):
- Stanford University Cancer Institute, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Ixazomib (MLN9708): Participants receive ixazomib (orally) PO on days 1, 4, 8, and 11. Treatment repeats every 21 days for up to 12 courses in the absence of disease progression or unacceptable toxicity.
Period: Overall Study
Arm/Group | Ixazomib (MLN9708)
Started | 4
Completed | 2
Not Completed | 2
Not completed — Withdrawal by Subject | 1
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Arm/Group | Ixazomib (MLN9708)
Number analyzed (Participants) | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 4
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 2
  More than one race | 0
  Unknown or Not Reported | 1

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate (ORR)
Description: Overall response rate after 3 cycles of treatment (9 weeks) was assessed as complete remission (CR); CR with incomplete recovery (CRi); and partial remission (PR) with MLN9708, in participants with NPM1-mutated AML by LeukemiaNet1 guidelines:
  Although achievement of complete remission (CR) has unique clinical significance for improved overall survival (OS) and relapse-free survival (RFS) compared to achievement of CRi with incomplete platelet recovery, the latter is still a clinically meaningful response, as it is independently-superior to resistant disease.
  Partial remission (PR) is defined as meeting all hematologic criteria for CR with an allowance for 5% to 25% bone marrow blasts or decrease of pre-treatment bone marrow blast percentage by at least 50%.
  Stable disease is defined as a change in bone marrow aspirate blast count within 10% of baseline.
  Relapsed disease is defined as reappearance of blasts in the blood or bone marrow blasts
Time Frame: 9 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Ixazomib (MLN9708)
Number analyzed (Participants) | 2
Participants
  Complete Remission (CR) | 0
  Complete Remission with incomplete recovery (CRi) | 0
  Partial Remission (PR) | 0
  Stable Disease (SD) | 0
  Relapsed Disease (RD) | 0
  Progressive Disease (PD) | 2

2. Secondary Outcome: Duration of Response (DOR)
Description: Duration of response (DOR) in participants with complete remission (CR) was defined as the period of time from documented complete remission through relapse or death, with relapse defined as reappearance of blasts in the blood or bone marrow blasts, after documented CR. DOR was to be assessed through at least 1 year follow-up.
Time Frame: 1 year
Population: No participants met the criteria of complete remission (CR), and so duration of response (DOR) in those participants could not be assessed.
Arm/Group | Ixazomib (MLN9708)
Number analyzed (Participants) | 0

3. Secondary Outcome: Overall Survival (OS)
Description: Overall survival (OS) from time of study entry to the earlier of death from any cause or end of follow up at 1 year
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Ixazomib (MLN9708)
Number analyzed (Participants) | 4
Participants | 0

4. Secondary Outcome: Serious Adverse Events Related to Ixazomib
Description: Ixazomib toxicity and tolerability were assessed based on the non-hematologic toxicities ≥ Grade 3 determined to be possibly, probably, or definitely related to the study agent Ixazomib.
  Adverse events that are possibly, probably, or definitely related to the study agent are considered "toxicities." The outcome is reported as the overall number of non-hematologic toxicities ≥ Grade 3.
Time Frame: 1 year
Population: All treated subjects are included.
Measure: Number; unit: Related adverse events
Arm/Group | Ixazomib (MLN9708)
Number analyzed (Participants) | 4
Related adverse events | 3

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Ixazomib (MLN9708)
All-Cause Mortality (participants affected / at risk) | 4/4
Serious Adverse Events (participants affected / at risk) | 4/4
Other Adverse Events (participants affected / at risk) | 4/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ixazomib (MLN9708) (N=4)
Febrile Neutropenia (Infections and infestations) | 1 (1)
AML Disease progression (Blood and lymphatic system disorders) | 2 (2)
Pancytopenia (Blood and lymphatic system disorders) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 2 (2)
Nausea (Gastrointestinal disorders) | 1 (1)
Dehydration (General disorders) | 1 (1)
Acute Respiratory Distress Syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Cardiopulmonary Arrest (Cardiac disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ixazomib (MLN9708) (N=4)
Acute Pulmonary Edema (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Skin Rash (Skin and subcutaneous tissue disorders) | 2 (2) — including: Maculo-papular rash
Vomiting (Gastrointestinal disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 2 (2)
Dysphagia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (2)
Rectal Pain (Renal and urinary disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No